CLINICAL TRIAL: NCT04519554
Title: Hysteroscopic Guided Endometrial Sampling: Prospective Comparison Between 5Fr and 7Fr Biopsy Forceps (HYSTEROBIO)
Acronym: HYSTEROBIO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: APHP200243; 2017-A00621-52 (Other: IDRCB)
Record Dates: First submitted 2020-08-17; First posted 2020-08-19 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Biopsy
Keywords: endometrial sampling hysteroscopy; postmenopausal bleeding; endometrial carcinoma
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5FR + 7FR (Other): Each woman is its own control and had biopsies with the 2 size of forceps. In this group first with 5FR then 7 FR
  Interventions: Device: Endometrial sampling
- 7FR + 5FR (Other): Each woman is its own control and had biopsies with the 2 size of forceps. In this group first with 7FR then 5FR
  Interventions: Device: Endometrial sampling

INTERVENTIONS:
Device: Endometrial sampling — Endometrial sampling with 2 different forceps

SUMMARY:
Indication for hysteroscopic guided biopsy compared to blind biopsy have been little evaluated. However, this kind of biopsy is usually performed in many centre. They allow exploration of uterine cavity but also to perform guided biopsies on the most suspicious area. However, with 5Fr forceps, biopsy are often too small to conclude.

DETAILED DESCRIPTION:
Blind biopsies using Novak or Cormier cannula had limits. Demirkiran et al conclude on 673 women that histology was similar between biopsies and hysterectomy in only 67% of cases. Others studies conclude thatit is difficult to conclude about focal disease with blind biopsies.

A study compared blind biopsies to biopsy performed under hysteroscopic guidance in women using Tamoxifene and conclude that guided biopsies were more specific (80% versus 68.9%) and a better positive predictive value (68.9% versus 43.7%) for all kind of endometrial pathologies

ELIGIBILITY:
Inclusion Criteria:

* • Woman over 18 year-old with abnormal uterine bleeding (or endometrium thickness over 10mm) and risk factors of endometrial carcinoma, or endometrium thickness over 5mm in a menopausal woman or abnormal uterine bleeding after 45 years old.

  * Woman who speak and understand french
  * Woman who give her written informed consent
  * Woman covered by french medical insurance

Exclusion Criteria:

* • Pregnant or breastfeeding patient

  * Patient under guardianship, curators or safeguard of justice.
  * Patient participating in another ongoing study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2020-09-20 (Estimated); Primary Completion 2021-12-20 (Estimated); Study Completion 2021-12-20 (Estimated)

PRIMARY OUTCOMES:
To evaluate ability to give a pathologic conclusion after 5Fr and 7Fr forceps biopsies | During the pathologist's analysis
  Evaluated by the number of cases on witch the biopsy allowed to conclude

SECONDARY OUTCOMES:
To compare histologic conclusions after 5 and 7Fr biopsies | During the pathologist's analysis
  Evaluated by Importance of collapse artifacts
To compare rate of ability to obtain pathologic conclusion on the sample after 5Fr and 7Fr forceps in endometrial carcinoma | During the pathologist's analysis
  The number of endometrial malignancies diagnosed histologically with either forceps
To evaluate the rate of hysteroscopic failure due to cervical stenosis | During the pathologist's analysis
  The number of cases where hysteroscopy was not possible

CONTACTS AND LOCATIONS:
Overall Officials: Perine CAPMAS, Principal Investigator — APHP
Locations (1):
- AP-HP, Bicêtre Hospital, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No